CLINICAL TRIAL: NCT00905047
Title: Open Comparative Study With a Cross-over According to Patients'Preference Receiving Xeloda or UFT With Folinic Acid in Advanced or Metastatic Colo-rectal Cancer
Brief Title: Xeloda or UFT (Tegafur-uracil) With Folinic Acid in Advanced or Metastatic Colorectal Cancer
Acronym: COLOCROSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: COLOCROSS
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Cancer
Keywords: colo-rectal cancer; advanced; metastatic; locally advanced or metastatic colo-rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Neoplasm Metastasis | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XELODA (Other)
  Interventions: Drug: XELODA
- UFT (Other)
  Interventions: Drug: TEGAFUR URACIL - FOLINIC ACID

INTERVENTIONS:
Drug: XELODA — XELODA, 2500 mg/m²/bid, with approximatively an interval of 12 hours, 30 minutes after breakfast and dinner - during 14 days.
  Cycle treatment duration : 21 days
  Arms: XELODA
Drug: TEGAFUR URACIL - FOLINIC ACID — Tegafur 300 mg/m2/tid with folinic acid 75 mg/tid during 28 days.
  Duration of treatment cycle : 35 days.
  Arms: UFT

SUMMARY:
The scope of the trial is to determine the preference of patients, after randomization and cross-over, for one of the two treatments.

Another objective of the trial is to assess and compare the safety of each treatment.

DETAILED DESCRIPTION:
Further study details as provided by Centre Oscar Lambret.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic colo-rectal cancer
* Age > or = 18 years old
* PS-WHO < or = 2
* Polynuclear neutrophil leukocytes > or = 1500/mm3, platelets > or = 100000/mm3
* Total bilirubin < or = 3 ULN, ASAT-ALAT < or = 2.5 ULN
* Effective contraception
* Written informed consent signed

Exclusion Criteria:

* Concomitant radiotherapy
* Contraindication to fluoropyrimidines
* Treatment with sorivudine and its chemical analogs such as brivudine
* Severe hepatic insufficiency
* Severe renal insufficiency
* Pregnant or lactating woman
* Hypersensitivity to capecitabine, 5FU, tegafur or one of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-09; Primary Completion 2010-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
patients preference after randomization and cross-over | after 2 cycles of treatment

SECONDARY OUTCOMES:
safety of each treatment | at day 56 (after two cycles of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: ADENIS Antoine, MD,PhD, Principal Investigator — Centre Oscar Lambret
Locations (13):
- France (13):
  - Centre Paul Papin, Angers
  - Centre Hospitalier, Armentières
  - Centre Hospitalier de Béthune, Beuvry
  - Centre Hospitalier de CHOLET, Cholet
  - Centre Leonard de Vinci, Dechy
  - Polyclinique du Bois, Lille
  - Centre Oscar Lambret, Lille
  - Hopital Saint Vincent de Paul, Lille
  - Centre Hospitalier Regional, Lille
  - Centre Hospitalier, Roubaix
  - Centre Joliot-Curie, Saint Martin Les Boulogne
  - Centre Hospitalier, Valenciennes
  - Clinique des Dentellieres, Valenciennes